CLINICAL TRIAL: NCT07387081
Title: An Open-label, Multicenter Phase II Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of LM-24C5 in Combination With Other Anti-tumor Treatment in Subjects With CEACAM5-positive Advanced Solid Tumors
Brief Title: Phase II Study of LM-24C5
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM24C5-02-201
Record Dates: First submitted 2025-12-02; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-24C5 in combination with anti-tumor therapies (Experimental)
  Interventions: Drug: LM-24C5
- LM-24C5 in combination with other anti-tumor therapies (Experimental)
  Interventions: Drug: LM-24C5

INTERVENTIONS:
Drug: LM-24C5 — Q2W Administered intravenously Drug: Penpulimab Q2W Administered intravenously Drug: Docetaxel Q3W Administered intravenously
  Arms: LM-24C5 in combination with anti-tumor therapies
Drug: LM-24C5 — Q2W Administered intravenously Drug: Penpulimab Q2W Administered intravenously Drug:Trifluridine and Tipiracil Hydrochloride Tablets BID,Oral Administration Drug:Bevacizumab Injection Q2W Administered intravenously
  Arms: LM-24C5 in combination with other anti-tumor therapies

SUMMARY:
This study is to evaluate the efficacy and safety of the LM-24C5 in combination with other therapies in subjects with CEACAM5-positive advanced solid tumor

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged 18-80 years old (including boundary values) , male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, or currently lack or are intolerant of, standard therapy.
6. CEACAM5-positive subjects.
7. At least one evaluable lesion.
8. Subjects must show appropriate organ and marrow function inlaboratory examinations within 7 days prior to the first dose.
9. Subjects who can communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Subjects with a history of other malignancies within 5 years prior to first dosing of LM-24C5, excluding cured squamous cell carcinoma of the skin, basal cell carcinoma, non-muscle-invasive bladder cancer, or localized low-risk prostate cancer, carcinoma in situ of the cervix/breast, and other malignancies deemed by the investigator to potentially benefit from participation in this study.
2. Subjects who have received other anti-tumor treatments before the first dosing of LM-24C5.
3. Previous immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis.
4. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
5. Present peripheral sensory or motor neuropathy ≥ grade 2.
6. Subjects with uncontrolled pain.
7. Subjects with symptomatic and untreated central nervous system metastases, and/or meningeal metastases.
8. Subjects who have uncontrollable third space effusion.
9. Previously received targeted therapy for same target.
10. . Use of any live vaccines within 28 days prior to 1st dosing of IMP.
11. Subjects with current or previous interstitial lung diseases or pneumonia requiring oral or intravenous glucocorticoids for adjuvant therapy.
12. Subjects on anticoagulants, such as heparin and vitamin K antagonists.
13. Clinically uncontrollable persistent recurrent vomiting.
14. Uncontrollable/severe gastrointestinal bleeding, ulceration or diarrhea within 28 days prior to first dose of IMP.
15. Subjects who received major surgery or interventional treatment within 28 days prior to the first dosing of IMP.
16. Subjects who have severe cardiovascular disease.
17. Subjects who have uncontrolled or severe illness.
18. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of IMP.
19. Subjects with a known history of autoimmune diseases.
20. Subjects who have a history of immunodeficiency disease.
21. Subjects with HIV infection, active HBV or HCV infection.
22. Child-bearing potential female who have positive results in pregnancy. test within 7 days before the first dose or are lactating.
23. Subject who have a known psychiatric diseases or disorders that may affect compliance with the trial.
24. Subject who is judged as not eligible to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-05-21 (Estimated); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
ORR | 110weeks
  Objective response rate

SECONDARY OUTCOMES:
Anti-tumor Activity | 110weeks
  Based on RECIST v1.1, evaluated progression-free survival (PFS), duration of response (DOR), disease control rate (DCR = CR + PR + SD), and change in target lesions relative to baseline; overall survival (OS).
PK Parameter（AUClast） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
Immunogenicity of LM-24C5 | baseline and 110 weeks
  ADA、Nab
Correlation between CEACAM5 and/or PD-L1 expression levels and treatment efficacy. | baseline and 110 weeks
  Correlation between CEACAM5 and/or PD-L1 expression levels and treatment efficacy.
PK Parameter（AUCtau） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Cmax） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Tmax） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（T1/2） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（ss） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Cmin） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（CLss） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Vss） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Rac） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（AUC） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Cmax, DF, etc.
PK Parameter（Cmax） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Rac, Cmax, DF, etc.
PK Parameter（DF） | baseline and 110 weeks
  Including but not limited to AUClast, AUCtau, Cmax, Tmax, T1/2, Cmax, ss, Cmin, ss, CLss, Vss, Rac, AUC, Rac, Rac, Cmax, DF, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Shanghai East Hospital, Shanghai, Shanghai Municipality